Official Title: Enhancing Older Adults' Everyday Memory Function

NCT Number: NCT04088136

Document Date: June 24, 2021

## Georgia Institute of Technology School of Psychology Christopher Hertzog, Principal Investigator Ann Pearman, Co-Investigator

## **Enhancing Older Adults' Everyday Memory Function**

## Key Information for Study 2 To be read prior to Consent Form

\*Of note, during the COVID-19 social distancing period, this program will only be offeredonline. We will use a Zoom meeting platform with password protected sessions.\*

#### What am I being asked to do?

You are being asked to be a volunteer in a research study. This page will give you key information to help you decide if you would like to participate. Your participation of voluntary. As you read, please feel free to ask any questions you may have about the research.

#### What is this study about and what procedures will you be asked to follow?

The purpose of this study is to see if different types of memory training can help older adults with everyday functioning. First, you will be asked to attend a virtual session where you will complete an intake interview over the phone and then engage in some pretest forms over your computer. Then, you will take part in one of two types of memory courses, which last three hours per day for four days over the course of 2 weeks. Following the memory courses, you will be asked to participate in one week of coaching, where you will be regularly contacted over the telephone by the research team. During this time, you will also record when you have a memory issue or success using a smartphone provided by the research team. You will also receive random prompts about your memory on the smartphone. Following the coaching week, you will continue reporting on your daily experiences for one more week. Finally, you will complete post-testing and return all provided equipment. Data collected from you during this study include information about your memory and mood, daily reports of your memory function, and interview information about your habits and routines. Your participation in this study is expected to last approximately 35-40 hours over the course of six to eight weeks.

# Are there any risks or discomforts you might experience by being in this study?

There is minimal risk for taking part in this study other than those involved in day to day life other than those involved in daily activities such as taking a class, keeping a calendar, or using a Smartphone. If you already carry a Smartphone, you'll have to carry a second phone with you which you might find cumbersome. You might get bored or annoyed with answering questions multiple times a day. You will never be required to answer questions you do not want to answer or take part in an activity in class or other times you do not want. You may quit the study at any time. There are no costs toyou other than your time.

## What are the reasons you might want to volunteer for this study?

The benefits of taking part in this study include contributing to the science of memory training in older adults as well as possibly improving your everyday memory functioningor learning new memory techniques.

You will be compensated for each completed step of this study. As compensation foryour time, we are offering payment up to \$190.

## Do you have to take part in this study?

It is fully your decision if you wish to be in this study or not. If you choose not to participate, or choose to participate and later determine you no longer wish to, you willnot lose any rights, services, or benefits as a result of your withdrawal. The study is completely voluntary.

## Georgia Institute of Technology School of Psychology Christopher Hertzog, Principal Investigator Ann Pearman, Co-Investigator

#### **Enhancing Older Adults' Everyday Memory Function**

## **Consent Form for Study 2**

#### **Introduction:**

You are being asked to take part in a research study. This intervention study is designed to investigate two different types of memory training procedures. There are no serious risks to participating in this study, however, it will take approximately 35-40hours of your time.

## Purpose:

This purpose of this study is to compare two types of memory training to see which, ifeither, is most effective for improving everyday functioning.

#### **Inclusion Criteria:**

The inclusion criteria are (1) access to the internet by phone or computer, (2) between 70 and 85 years of age, (3) English-speaking, (4) identify as in fair to good health, (5) no diagnosed illness that can cause impairment in cognitive functioning (e.g. Alzheimer's disease or vascular dementia), and (6) located in the US during the time of participation.

#### **Exclusion Criteria:**

The exclusion criteria are (1) no access to internet, (2) not between 70 and 85 years of age, (3) non-English-speaking, (4) in poor health, (5) diagnosed illness that can cause cognitive impairment, and (6) located in non-US country.

#### **Procedures:**

There are several parts to this study. The total time required will be about 35 – 40hours.

The first part of the study is a virtual meeting with an intake interview on Zoom and the pretest which will be done online. After these, you will be assigned to either an everyday skills group or a memory strategy training group. This assignment will be random with the constraint that we end with equal numbers of people in both groups. Regardless of the group in which you are assigned, you will be asked to attend four in-person intervention sessions online. These sessions will be three hours in length and will be held over two weeks. You will

be assigned briefhomework assignments as well as check-in calls from the staff after the first three sessions of the intervention. During this time you will also be sent a loaner phone and you will be trained to use it.

Once the courses are over, participants enter a one week coaching program. During this time, you will be encouraged to practice the skills you learned in the course. In addition, we will also ask you to fill out daily forms about your memory experiences each day and you will be prompted on the Smartphone to answer some questions several times a day as well as filling out some forms each night. In total, these questions will take about 45 – 60 minutes/day. This one-week period includes additional phone contacts with a member of the research team to discuss and coach your use of the memory skills and to check-in with you to see how things are going. These calls are designed to help you really "get" the techniques we taught. Both groupswill have similar amounts of phone contact and homework during this time.

Once the coaching week is complete, you would enter a measurement period which will last for one week. During this time, we would ask you to continue doing the daily diaries, phone prompts and recording, and memory questions. This will take about 45 –60 minutes per day.

The final part of this study will involve an online posttest. This will allow us to evaluate the program as well as to investigate potential improvements in program administration. During this session, you will also be asked to mail the loaner Smartphone back to the lab. You will be debriefed at the end of this session.

Your time commitment for this study will be as follows:

- 1) Virtual interview, questionnaires, and pretest: 3-4 hours
- 2) Intervention Sessions: 4 virtual classes for 3 hours/class over the course of one week + 3 nights of homework and phone calls (30 minutes each)
- 3) One-week of coaching and homework: 5-7 hours over the course of 1 week
- 4) One-week additional measurement period: 45-60 minutes/day for one week
- 5) Online posttest: 3 hours

The total time for the study will be about 35 - 40 hours.

#### **Risks or Discomforts:**

There is minimal potential risk for taking part in this study other than those involved in daily activities such as taking an online class, keeping a calendar, or talking on the phone. You might find it inconvenient to carry a second phone. You will never be required to answer questions you do not want to answer or take part in an activity in class that you do not want. You may quit the study at any time. There are no costs to you other than your time.

#### **Benefits:**

There is potential for you to benefit from this study. Both techniques we will be teaching have a history of being effective in helping people feel better about their memory. Also, we hope to take the information we learn from you and expand the study to include more people. For this, we will also ask questions at the end about what you thought

about the study and what can be improved as a way of benefiting future studies. Your opinions and thoughts will be extremely valuable to us.

## **Compensation to You:**

You will be compensated for taking part in each part of this study as follows:

- 1) Completion of in-person interview, questionnaire & pretest: \$25
- 2) Completion of four intervention classes (\$10/session): \$40
- 3) One-week coaching period: (\$5/day) \$35
- 4) One-week measurement period: (\$10/day) \$70
- 5) Completion of in-person interview & posttest: \$20

If you stop taking part in the study at any point, you will only be compensated forcompleted sessions.

U.S. Tax Law requires that a 1099-misc be issued if U.S. tax residents receive \$600 or more per calendar year. If non-U.S. tax residents receive more than \$75, mandatory 30% withholding is required. Your address and citizenship/visa status and tax I.D. maybe collected for compensation purposes only. This information will be shared only withthe Georgia Tech department that issues compensation for your participation.

#### **Storing and Sharing your Information:**

Your participation in this study is gratefully acknowledged. It is possible that your information/data will be enormously valuable for other research purposes. By signing below, you consent for your de-identified information/data to be stored by the researcher and to be shared with other researchers in future studies. If you agree to allow such future sharing and use, your identity will be completely separated from your information/data. Future researchers will not have a way to identify you or to link your responses to your name. Any future research using your data must be approved by an ethics committee before beingundertaken.

#### **Confidentiality:**

The following procedures will be followed to keep your personal information confidential in this study:

- We will comply with any applicable laws and regulations regarding confidentiality.
- To protect your privacy, your records will be kept under an identification number rather than by your actual name.
- The records will be kept in locked files or in encrypted files and only authorized research and staff will be allowed to look at them.
- Your name and any other fact that might point to you will not appear when results of this study are presented or published.
- You should be aware that when the study is conducted in an online formatit
  will not be run from a secure https server of the kind typically used to
  handle credit card transactions, so there is a small possibility that an
  unauthorized third party may interfere with our sessions. However, weuse
  password protected sessions to minimize the likelihood of this.

• To make sure this research is carried out in the proper way, the Georgia Institute of Technology IRB and the Office of Human Research Protections may look over study records during required reviews.

## **ClinicalTrials.gov**:

A description of this study will be available on http://www.ClinicalTrials.gov, as requiredby U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Additional guidance, including the definition of <u>clinical trials</u>, may be found at www.researchintegrity.gatech.edu.

#### **Questions about the Study:**

You may contact Dr. Christopher Hertzog with questions. Phone:

404-894-6774

Email: <a href="mailto:christopher.hertzog@psych.gatech.edu">christopher.hertzog@psych.gatech.edu</a>

#### In Case of Injury/Harm or Adverse Reactions:

Although we do not anticipate any harm because of taking part in this study, reports ofinjury or reaction should be made to PI Christopher Herzog, Ph.D., at 404-894-6774. Neither the PI nor Georgia Institute of Technology has made provision for payment of costs associated with any injury resulting from participation in this study.

#### **Questions about Your Rights as a Research Participant:**

- Your participation in this study is voluntary. You do not have to be in this study if you don't want to be.
- You have the right to change your mind and leave the study at any time without giving any reason and without penalty.
- Any new information that may make you change your mind about being in this study will be given to you.
- You will be given a copy of this consent form to keep.
- You do not waive any of your legal rights by signing this consent form.

If you have any questions about your rights as a research participant, you may contact Ms. Kelly Winn, Georgia Institute of Technology Office of Research Integrity Assurance, at (404) 385- 2175.

For this consent form, we are using a "virtual signature". Signing your name in the

| box below will indicate that you have re information given in this consent form, a study. | | • |
|---|---|---|
| Participant Name (printed) | Participant Signature | Date |
| Signature of Person Obtaining Consent | <br>Date | |

# **Consent to Store and Share your Information:**

# Please choose one of the following:

| $oldsymbol{\Theta}$ I agree that my de-identified information/data may be stored and shared for future unspecified research. |
|---|
| Initials |
| $oldsymbol{\Theta}$ I do not allow my de-identified information/data to be stored and shared for future, unspecified research. These may only be used for this specific study. |
| Initials |